CLINICAL TRIAL: NCT00120172
Title: A Phase II Study of Oxaliplatin, Capecitabine, and Bevacizumab in the Treatment of Elderly Patients With Metastatic Colorectal Cancer
Brief Title: Study of Oxaliplatin, Capecitabine, and Bevacizumab to Treat Older Patients With Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: positive results from a larger study with same regimen was released.
Sponsor: Geriatric Oncology Consortium (Other)
Collaborators: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOC-GI-010
Record Dates: First submitted 2005-07-08; First posted 2005-07-15 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Colorectal Cancer; Neoplasm Metastasis
Keywords: colorectal; metastatic; elderly; metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Oxaliplatin; Capecitabine; Bevacizumab

INTERVENTIONS:
Drug: oxaliplatin, capecitabine, bevacizumab

SUMMARY:
Currently there is no one standard of care for older patients with metastatic colorectal cancer. The study will examine the tumor response to capecitabine, oxaliplatin, plus bevacizumab. The study will also gather information on the usefulness and side effects of this treatment combination.

DETAILED DESCRIPTION:
Colorectal cancer is primarily a disease of the elderly, with the median age in the United States of 70 years. Age greater than 65 years at presentation is not a contraindication to standard therapies; acceptable morbidity and mortality, as well as long term survival, are achieved in this patient population. However, studies evaluating combination therapy have generally involved younger patients with high performance status scores. Given the non-over-lapping safety profiles of the proposed study agents and the potential synergy, it would be of benefit to explore the combination of oxaliplatin, capecitabine, and bevacizumab in the treatment of older patients with colorectal cancer. Time to progression, overall response, duration of response, and toxicity profile will be evaluated. The feasibility of using a self-report geriatric assessment tool will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years and above;
* Histologically or cytologically documented adenocarcinoma of the colon or rectum;
* Metastatic disease;
* Measurable disease or assessable but nonmeasurable disease allowed;
* ECOG 0-1
* No prior oxaliplatin or bevacizumab.
* No prior chemotherapy for metastatic disease. Prior adjuvant chemotherapy allowed;
* No prior fluoropyrimidine therapy (unless give in an adjuvant setting and completed at least 4 months earlier);
* No bleeding diathesis or coagulopathy
* Adequate renal and hepatic functions as per protocol;
* Signed informed consent

Exclusion Criteria:

* Clinically significant cardiovascular or peripheral vascular disease;
* Concurrent chronic aspirin, nonsteroidal anti-inflammatory drugs, warfarin, or therapeutic heparin;
* Serious non-healing wound, ulcer, or bone fracture;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy (measured by time to progression) of oxaliplatin, capecitabine, and bevacizumab as first-line therapy in elderly patients with metastatic colorectal cancer.

SECONDARY OUTCOMES:
Overall response
Duration of response
Safety and tolerability (NCI CTCAE v3.0, discontinuations, dose intensity)
Vulnerable Elders Survey (VES-13) and Geriatric Depression Scale (GDS) scores

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Lichtman, MD, Study Chair — Geriatric Oncology Consortium
Locations (5):
- United States (5):
  - Mission Hills, California
  - Washington D.C., District of Columbia
  - Inverness, Florida
  - New Port Richey, Florida
  - Coeur d'Alene, Idaho